CLINICAL TRIAL: NCT06507228
Title: North West London Pebble Pathway: Automated OSA Diagnosis
Acronym: PEBBLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patrik Bachtiger (Other)
Responsible Party: Sponsor-Investigator, Patrik Bachtiger, NIHR Academic Clinical Lecturer, Imperial College London
Organization: Imperial College London (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA8366
Record Dates: First submitted 2024-07-06; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Propspective real world implementation and health economic study; historical control group for comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NWL PEBBLE STT patients (Other): Real-world clinical care arm investigating novel pathway
  Interventions: Diagnostic Test: NWL PEBBLE STT

INTERVENTIONS:
Diagnostic Test: NWL PEBBLE STT — At home testing for OSA with AcuPebble.

SUMMARY:
Patients with obstructive sleep apnoea (OSA) wait up to two years for a diagnostic test. Early diagnosis enables optimal treatment, mitigating risks including heart failure, lung disease, and stroke. Current diagnostic approaches are expensive (£391), time-consuming (>1-hour interpretation), uncomfortable (cables/tubes/wires), and inequitable (multiple hospital visits). Overcoming all these limitations, we have designed and will investigate a straigh-to-test automated diagnostic pathway for OSA. This will use the AcuPebble, a miniature wearable acoustic sensor and the first regulated technology for automated, at-home diagnosis. The test is cheap (< £100); time-saving; endorsed by patients, and accessible (posted directly to patients). This project will measure the impact of a potentially transformative, innovative, and scalable diagnostic pathway using AcuPebble technology.

DETAILED DESCRIPTION:
The investigators are conducting a prospective implementation and health economic study of a novel straight-to-test (STT) clinical diagnostic pathway for OSA, using a novel, regulatory-approved wearable medical device for automated diagnosis of OSA in the home setting (AcuPebble SA100). The setting is real-world direct clinical care, with participation from three NHS sleep medicine centres servicing the North West London region.

Inclusion criteria is primary care referrals for OSA investigation were triaged onto the pathway based on predetermined criteria, compared to a historical cohort of patients undergoing STT using cardiorespiratory polygraphy (CR-PG) technology serving as a control group. The primary outcome is time-to-diagnosis. Secondary outcomes include NHS cost-saving per patient; surrogates for health equity (e.g. test completion rates, time/cost of journeys saved); and carbon footprint reduction from averted patient journeys (sustainability).

ELIGIBILITY:
Inclusion Criteria:

* OSA testing referral from primary care

Exclusion Criteria:

* Unable to follow test instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis | 12 months
  Time to diagnosis vs. historical control group

SECONDARY OUTCOMES:
Cost saving per test | 12 months
  Cost saving per test in pounds sterling compared to control group
Test completion rate | 12 months
  Completion rate as proxy for health equity
Financial saving to patients from cutting journeys associated with appointments | 12 months
  Cost saved from averted journeys by per patient cost of public transport and time taken to travel; informed by mapping journey per patient post-code to sleep study centre.
Sustainability impacts by carbon footprint reduction | 12 months
  CO2 footprint from averted technologies (reduced plastic waste) and reduced patient journeys (CO2 footprint reduction from miles travelled, calculated using Echochain carbon footprint calculator).
Time saving to patients from cutting journeys associated with appointments | 12 months
  Time saved from averted journeys by per patient cost of public transport and time taken to travel; informed by mapping journey per patient post-code to sleep study centre.

CONTACTS AND LOCATIONS:
Locations (1):
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Sharable upon reasonable request.

REFERENCES:
- [Background] Devani N, Pramono RXA, Imtiaz SA, Bowyer S, Rodriguez-Villegas E, Mandal S. Accuracy and usability of AcuPebble SA100 for automated diagnosis of obstructive sleep apnoea in the home environment setting: an evaluation study. BMJ Open. 2021 Dec 21;11(12):e046803. doi: 10.1136/bmjopen-2020-046803. PMID 34933855